CLINICAL TRIAL: NCT06049953
Title: Developmental Effects of Antenatal Exposure to Antipsychotics
Brief Title: Maternal And Infant Antipsychotic Study
Acronym: MAIA
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Erasmus Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thalia Robakis, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY 23-00239; R01HD111117-01 (NIH)
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Antipsychotics; Pregnancy
Keywords: antipsychotic; pregnancy; severe mental illness; neonatal adaptation syndrome; neurodevelopment
MeSH Terms: conditions — Mental Disorders | interventions — Antipsychotic Agents; Antidepressive Agents; Benzodiazepines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paired whole blood and plasma samples obtained from the mother and from the umbilical cord at delivery will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Antipsychotic medication: Pregnant women with severe mental illness (diagnosis of bipolar disorder, primary psychotic disorder, or any history of psychiatric hospitalization) who are treated with any of the following medications during pregnancy: Quetiapine, olanzapine, risperidone, aripiprazole, ziprasidone, lurasidone, haloperidol, or any other medication in the first- or second-generation antipsychotic class. All orally administered, with dosages titrated to clinical effect by the participant's primary psychiatrist.
  Interventions: Drug: Antipsychotics
- Non-antipsychotic medication: Pregnant women with severe mental illness (diagnosis of bipolar disorder, primary psychotic disorder, or any history of psychiatric hospitalization) who are treated with any psychotropic medications during pregnancy other than those listed.
  Interventions: Drug: Non-antipsychotic medication
- No medication: Pregnant women with severe mental illness (diagnosis of bipolar disorder, primary psychotic disorder, or any history of psychiatric hospitalization) who are not treated with any psychotropic medications during pregnancy.
  Interventions: Other: No Medication

INTERVENTIONS:
Drug: Antipsychotics — Antipsychotic medications are widely prescribed for severe mental illness such as affective and non-affective psychosis, mood stabilization, and augmentation of unipolar depression.
  Groups: Antipsychotic medication
Drug: Non-antipsychotic medication — Psychotropic medications are typically prescribed to manage symptoms of anxiety, depression, psychological distress, and/or insomnia.
  Other Names: Antidepressants; Benzodiazepines
  Groups: Non-antipsychotic medication
Other: No Medication — Non-psychotropic medications
  Groups: No medication

SUMMARY:
The goal of this observational study is to learn about maternal psychiatric course and infant development in pregnant individuals with severe mental illness, comparing those treated with antipsychotics to those treated with other medications or without medication. The main questions it aims to answer are:

1. Is risk of psychiatric relapse different among individuals who take antipsychotic medication, other medication, or no medication?
2. Are pregnancy and neonatal health outcomes different among individuals who take antipsychotic medication, other medication, or no medication?
3. Do infant behavior and neurodevelopment differ among babies who were exposed to antipsychotic medication, other medication, or no medication in utero? Participants will

   * complete a psychiatric interview and questionnaires while pregnant;
   * donate blood from the mother and from the umbilical cord at delivery
   * have their babies participate in infant behavior evaluations and an EEG procedure.

Researchers will compare these outcomes among individuals who were treated either with antipsychotic medication, with psychotropic medications of other classes, and with no medication, to see if psychiatric benefits for the mother and health outcomes for mother and child differ among these three types of treatment.

DETAILED DESCRIPTION:
Antipsychotic (AP) medications are widely prescribed for a range of mental illnesses including bipolar disorder and nonaffective psychosis. These disorders usually onset in adolescence or early adulthood; thus, women of childbearing age are among those prescribed APs. The number of pregnancies exposed to APs has been increasing over time. Yet their efficacy has never been definitively demonstrated in this population.

APs cross the placenta and block dopamine (DA) D2 receptors, which are functional in the developing fetus, including influencing the proliferation and differentiation of neural progenitor cells. Increased DA signaling in early development results in increased numbers of inhibitory cortical interneurons and decreased numbers of pyramidal cells, while decreased DA signaling has the reverse effect. Thus, tonic DA blockade in utero could alter the excitatory/inhibitory balance in mature prefrontal cortex, which could affect fear processing, social functioning, and spatial or working memory in the long term. Additionally, gestational diabetes mellitus (GDM) is an established short-term risk of AP in pregnancy, which is associated with both increased body size and impaired cognitive and motor development in offspring.

At present very limited data exist on developmental outcomes associated with antenatal exposure to APs. Infant studies have found some evidence of initial difficulty adapting to life outside the womb as well as early neuromotor problems, but existing studies lack adequate comparison groups, and longitudinal data are lacking. Regarding long-term outcomes, the research group has found sex-specific increases in risk for psychiatric disorders for male, but not female, offspring, in both a register-based dataset and a clinical pilot study. This potential neurodevelopmental vulnerability requires further investigation in a rigorous longitudinal cohort study.

This study aims to investigate efficacy and adverse effects of AP exposure in pregnant women with severe mental illness (SMI). The research team hypothesizes that APs will be efficacious for psychiatric disorders, but will be associated with increased weight gain in mothers, poor neonatal adaptation in neonates, and sex-specific neurodevelopmental changes in infants. The overall goal is to precisely describe the risk/benefit ratio associated with AP treatment in pregnancy, in order to allow pregnant women with SMI to make informed decisions about their care.

Study Aims:

Aim 1: To investigate efficacy and adverse effects of AP treatment for pregnant women.

Aim 1a: Efficacy of AP treatment for pregnant women with SMI. Hypothesis: Women taking either APs or non-AP mood stabilizers will be less likely to relapse with mood or psychotic episodes than those not medicated.

Aim 1b: Adverse pregnancy outcomes with AP treatment for pregnant women. Hypothesis: Women taking APs will have greater weight gain in pregnancy than women taking non-APs or women taking no medication.

Researchers will recruit women in pregnancy with SMI (bipolar or primary psychotic disorder, N=200) in three groups: taking AP, taking other psychotropic medication, and taking no psychotropic medication, via two specialized perinatal psychiatric centers in NYC and the Netherlands. Women will be followed naturalistically and assessed for psychiatric relapse in pregnancy and the postpartum period, as well as complications of pregnancy, including weight gain and gestational diabetes, This will be the first study of AP efficacy in pregnancy.

Aim 2: To describe neonatal adaptation and physical growth in neonates of the mothers either exposed or unexposed to APs during pregnancy. Aim 2a: Neonatal adaptation in neonates either exposed or unexposed to APs during pregnancy. Hypothesis: Neonates of mothers who took APs during pregnancy will evince poorer neonatal adaptation than neonates of mothers who took either non-AP psychotropics or no medication. Aim 2b: Physical growth in neonates either exposed or unexposed to APs during pregnancy. Hypothesis: Neonates of mothers who took APs during pregnancy will have larger body sizes than neonates of mothers who took either non-AP psychotropics or no medication. The research team will examine obstetric and neonatal outcomes of infants of women with SMI, including neonatal adaptation syndrome (NAS), with control for maternal diagnosis and level of functioning. This will be the first controlled study of NAS after antenatal AP exposure.

Aim 3: To describe neurobehavioral development through 6 months in children from Aim 2. Aim 3a: Auditory sensory gating in children exposed to AP antenatally. Hypothesis: All infants prenatally exposed to APs will have reduced inhibitory activity as measured by the P50 component in the EEG. Aim 3b (Exploratory): Neurobehavioral development through 6 months in children exposed to AP antenatally. Hypothesis: Researchers predict increased symptoms of anxiety and internalizing behaviors for males only. Reduced auditory sensory gating will mediate, and sex will moderate, socioemotional outcomes associated with AP exposure. Comprehensive interviews, behavioral observations, and electroencephalography (EEG) obtained in a home visit at 6 months will assess socioemotional, cognitive, and motor development. The research team will investigate whether infant sex moderates any observed effects of AP exposure. This will be the first study of neural activity after antenatal AP exposure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Severe mental illness, including:

  * Psychotic disorder (affective and nonaffective)
  * Bipolar disorder
  * History of psychiatric hospitalization, regardless of diagnosis
* Able to complete study interviews and measures in English, Dutch, or Spanish

Exclusion Criteria:

* Active substance use disorder in pregnancy
* Insufficiently high-functioning to provide full informed consent and/or participate in study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with severe mental illness as defined in Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Mini-International Neuropsychiatric Interview | through study completion, an average of 6 months postpartum
  In the DSM-5 Mini-International Neuropsychiatric Interview (M.I.N.I.) researchers will conduct modules for major depressive episode, (hypo)manic episode, and psychotic disorders. A clinical structured interview with very precise questions about psychological problems will require a 'yes' or 'no' answer. The M.I.N.I. is divided into modules identified by letters, each corresponding to a diagnostic category. At the beginning of each diagnostic module (except for psychotic disorders module), screening questions(s) corresponding to the main criteria of the disorder are presented in a gray box. At the end of each module, diagnostic box(es) permit the clinician to indicate whether diagnostic criteria are met.
Finnegan Neonatal Abstinence Scoring System | 24 hours postnatal
  Symptoms of poor neonatal adaptation, as assessed by Finnegan scale at 24 hours of life. Finnegan Neonatal Abstinence Scoring System (NAS) is an observer-rated scale documenting signs of neonatal adaptation. The individual NAS symptoms are weighted (numerically scoring 1-5) depending on the symptom, and the severity of the symptom expressed. The total score ranges from 0 to 43. Infants scoring an 8 or greater are recommended to receive pharmacologic therapy.
Ratio of auditory evoked potentials as measured by EEG | 6 months postnatal
  Electrical activity of brain cells in response to a sound stimulus, measured noninvasively on the outside of the scalp by electroencephalography

SECONDARY OUTCOMES:
Maternal weight gain | through delivery, approximately 40 weeks post conception
  Total pregnancy weight gain
Oral glucose tolerance test score | at 24 weeks
  A glucose screening test is a routine test during pregnancy that checks a pregnant woman's blood glucose (sugar) level. Score on oral glucose tolerance test will be recorded.
Fetal body size | at 20 weeks
  Fetal ultrasound-based and infant anthropometric measurements
Fetal weight | at 20 weeks
Fetal head circumference | at 20 weeks
Fetal biparietal diameter | at 20 weeks
Fetal cerebellar diameter | at 20 weeks
Neonatal birth weight adjusted for gestational age at delivery, as a percentile score | at 20 weeks
Fetal femur length | at 20 weeks
Neonatal body size | at delivery
Neonatal length | at delivery
Neonatal weight | at delivery
Neonatal head circumference | at delivery
Changes in Infant length percentile | at delivery and 6 months postnatal
Changes in weight percentile | at delivery and 6 months postnatal
Bayley-III Score | at 6 months postnatal
  Neurodevelopmental assessment scores are age dependent and based motor and behavioral abilities, often reported for normal or abnormal for age. Bayley Scales of Infant and Toddler Development, third edition, (Bayley III) is an instrument designed to measure the developmental functioning of infants and toddlers between the ages of 1 month and 42 months (age adjustments for prematurity are accommodated with the tool). It provides age specific composite scores for cognitive (91 items, score min 55 max 145), language (98 items, score min 47 max 153), and motor (138 items, score min 46 max 154) skills. For all scales, higher scores indicate favorable outcomes and lower scores indicate possible delay/deficit.
Vineland Interview | at 6 months postnatal
  Socioemotional, cognitive, and motor development as measured by Vineland interviews. . The Vineland measures five domains: Communication, Daily Living Skills, Socialisation, Motor Skills, and Maladaptive Behaviour. Each domain is summed, and the domain scores are converted to standardized scores. The normative score is 100, with standard deviation of 15. A higher score (above 100) means better adaptive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Thalia Robakis, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored and shared in accordance with HIPAA and GDPR law. Deidentified data will be shared between the two sites for the purpose of analysis of study outcomes.
  For this purpose:
  * dataset will be deidentified
  * datasets will be limited
  * data will be aggregated
  * no directly traceable data will be shared
  * data keys will never be shared between sites
  * data will be encrypted
  The process will be legally supported by Data transfer Agreements.
  Deidentified US data will be stored at the NICHD Data and Specimen Hub (DASH). Deidentified Dutch data will be stored at the electronic archives at the Erasmus MC. Repositories will be accessible for researchers of the MAIA study with the proper access rights, only